CLINICAL TRIAL: NCT00018551
Title: 3389 Colorectal Adenoma: Chemoprevention With Folic Acid
Brief Title: Chemoprevention With Folic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: ONCO-021-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Colon Cancer; Adenoma; Colonic Polyps
MeSH Terms: conditions — Colonic Neoplasms; Adenoma; Colonic Polyps | interventions — Folic Acid

INTERVENTIONS:
Drug: Folic Acid

SUMMARY:
Colorectal neoplasia is the second most common cancer in the United States and other Western countries with about 140,000 newly diagnosed cases per year in the United States with a mortality rate of about 40%. The identification of a specific natural or synthetic compound with the ability to reverse or suppress the process of colon carcinogenesis would have profound implication in the development of colorectal adenomas and their subsequent transformation to colon cancer. Furthermore, the establishment of a correlative relationship between biomarkers of cell proliferation, differentiation, apoptosis and adenoma recurrence would provide pivotal data required to elucidate cell signaling mechanisms in future colon cancer chemoprevention trials.

ELIGIBILITY:
Asymptomatic individuals from the age of 18 -80 years, undergoing clinically indicated colonoscopy for colon polyps noted on screening flexible sigmoidoscopy or as routine surveillance for a history of colon polyps, who are found to have at least one adenoma > 0.5cm will be eligible for entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1998-10; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs, Detroit, Michigan, United States